CLINICAL TRIAL: NCT02504788
Title: A Prospective Study of the Impact of Hippocampal Avoidance During Whole Brain Radiotherapy on Neurocognitive Function Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-4151B
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Brain Metastasis; Brain Metastases
Keywords: Whole Brain Radiotherapy (WBRT); Neurocognitive Functions (NCFs); Hippocampus; Hippocampus Sparing during Whole Brain Radiotherapy (HS-WBRT)
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hippocampal-sparing WBRT (Experimental): All studied patients should undergo a computed tomography (CT) simulation scan encompassing the entire head region with 1.25-mm slice thickness using a thermoplastic mask for immobilization. To achieve conformal hippocampal sparing during the delivery of whole brain radiation (WBRT), the technique of volumetric modulated arc therapy (VMAT) via Linac-based RapidArc®.In terms of dose prescription, a dose of 30 Gy in 12 fractions was prescribed to whole-brain planning target volume (PTV) if the role of RT was considered either adjuvant following craniotomy with tumor removal or therapeutic for treating oligometastatic brain disease.
  Interventions: Radiation: hippocampal-sparing WBRT

INTERVENTIONS:
Radiation: hippocampal-sparing WBRT

SUMMARY:
Whole brain radiotherapy (WBRT) has long been a practical and effective therapeutic modality for various settings of management in radiation oncology. For example, the indications for WBRT should include brain metastasis or metastases, the setting of prophylactic cranial irradiation (PCI) used mainly for patients with limited-stage small cell lung cancer, and even some patients with extensive-stage small cell lung cancer. The rationales for WBRT are essentially based on that it can target both microscopic and gross intracranial disease.

In addition to providing rapid alleviation of neurologic symptoms and enhanced intracranial disease control, WBRT might also prolong the time to develop neurocognitive function (NCF) decline. However, paradoxically NCF decline can also occur due to a sequel of WBRT. In terms of the time course of WBRT-induced NCF decline, it might vary considerably according to the specific domains which are selected to be measured. Early neurocognitive decline occurs within the first 1 - 4 months after WBRT for brain metastases. The domains of early neurocognitive decline principally involve verbal and short-term memory recall.

Since several decades ago, it has been understood that hippocampus plays an essential role in memory function. Not little evidence supports that radiation-induced damage to hippocampus should be strongly associated with NCF impairment. Furthermore, several studies have shown that isodose distribution in hippocampus is closely related to neurocognitive function in patients with benign or low-grade brain tumors. As a consequence, it is hypothesized that conformal hippocampal sparing during the course of WBRT (HS-WBRT) might provide significant preservation in terms of cognitive function.

This prospective cohort study aims to explore and evaluate the impact of the delivery of HS-WBRT on the pattern of NCF change and the extent of NCF decline in patients receiving prophylactic or therapeutic WBRT. As compared with previous related and relevant studies, it will also be investigated whether neurocognitive functional preservation can be achieved via the integration of hippocampal sparing with the course of WBRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically-confirmed non-hematopoietic malignancy who are referred for therapeutic or prophylactic WBRT
* Good performance status no worse than Eastern Cooperative Group (ECOG) of 2 or a general status of Karnofsky Score (KPS) at least 70 %
* The number and extent of brain metastatic lesions should be no more than three metastatic foci with a greatest diameter no more than 4 cm

Exclusion Criteria:

* Patients with MRI-identified metastasis within 5 mm perihippocampally
* Clinical suspicion of leptomeningeal spreading
* History of prior radiotherapy including stereotactic radiosurgery delivered to brain/head region for any reasons

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is delayed recall, as determined by the change/decline in verbal memory (WMS III- Word List score) from the baseline assessment to 4 months after the start of HS-WBRT. | 4 months after the start of HS-WBRT
  Neurocognitive assessment: including memory, executive functions, and psychomotor speed. This neurocognitive outcome was delayed recall, as determined by the change/decline in either verbal memory [Wechsler Memory Scale - 3rd edition (WMS III) - Word List score] or non-verbal memory (WMS III- Visual Reproduction score) from the baseline assessment to 4 months after the start of the course of WBRT with hippocampus sparing (HS-WBRT). Additionally, the follow-up of neurocognitive assessment will also be administered at 12 months and up to 18 months after the start of HS-WBRT.
The primary endpoint is delayed recall, as determined by the change/decline in non-verbal memory (WMS III- Visual Reproduction score) from the baseline assessment to 4 months after the start of HS-WBRT. | 4 months after the start of HS-WBRT
  Neurocognitive assessment: including memory, executive functions, and psychomotor speed. This neurocognitive outcome was delayed recall, as determined by the change/decline in either verbal memory [Wechsler Memory Scale - 3rd edition (WMS III) - Word List score] or non-verbal memory (WMS III- Visual Reproduction score) from the baseline assessment to 4 months after the start of the course of WBRT with hippocampus sparing (HS-WBRT). Additionally, the follow-up of neurocognitive assessment will also be administered at 12 months and up to 18 months after the start of HS-WBRT.

SECONDARY OUTCOMES:
Overall survival time, indicated by the time from the date of recruitment to the date of expiring | up to 18 months
The time from the date of recruitment to that of intracranial progression/failure noted on brain MRI or CT | up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin SY, Tsan DL, Chuang CC, Yang CC, Pai PC, Wang CL, Wu YM, Lee CC, Lin CH, Wei KC, Chou WC. Oncological Outcomes After Hippocampus-Sparing Whole-Brain Radiotherapy in Cancer Patients With Newly Diagnosed Brain Oligometastases: A Single-Arm Prospective Observational Cohort Study in Taiwan. Front Oncol. 2022 Jan 12;11:784635. doi: 10.3389/fonc.2021.784635. eCollection 2021. PMID 35096584
- [Derived] Tsai PF, Yang CC, Chuang CC, Huang TY, Wu YM, Pai PC, Tseng CK, Wu TH, Shen YL, Lin SY. Hippocampal dosimetry correlates with the change in neurocognitive function after hippocampal sparing during whole brain radiotherapy: a prospective study. Radiat Oncol. 2015 Dec 10;10:253. doi: 10.1186/s13014-015-0562-x. PMID 26654128